CLINICAL TRIAL: NCT01985958
Title: A Pilot Study to Evaluate Radiotherapy-Induced Ant-Tumor Immunity in Metastatic Carcinoma of the Pancreas
Brief Title: A Pilot Study to Evaluate Radiotherapy-Induced Anti-Tumor Immunity in Metastatic Carcinoma of the Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: UPCC 14213
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Histological or Cytological Diagnosis of Pancreatic Carcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): In this trial, we will deliver low-dose (8Gy in a single fraction) radiotherapy (SBRT or any other acceptable delivery method as determined by the treating physician) for palliation of symptoms in patients in whom it is clinically indicated. This dose is far lower than what has been used in the definitive settings described above. This is a safe dose, and is entirely consistent with the dose range used for routine palliation. Therefore, this trial does not involve an experimental intervention; the research aspect of this protocol is the evaluation of the immune response to clinically indicated palliative radiotherapy.
  Interventions: Device: Radiation therapy

INTERVENTIONS:
Device: Radiation therapy

SUMMARY:
Primary Objective: To estimate the rate at which radiotherapy to the primary or a metastatic lesion produces an immune response in patients with metastatic carcinoma of the pancreas.

Secondary Objectives: To characterize the kinetics of an immune response induced by radiotherapy. To characterize the dependency of the immune response on prior exposure to chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of pancreatic carcinoma
* Patients ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1,or 2
* Patients must have distant metastatic disease (stage 4)
* Satisfactory organ and bone marrow function as defined by: Absolute neutrophil count> 1,000/uL, Platelets > 75,000uL Hemoglobin > 9 Bilirubin ≤ 2.0x the institutional normal upper limit unless secondary to bile duct obstruction by tumor,
* Creatinine ≤ 1.5x the institutional normal upper limit
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5x the institutional normal upper limit.
* A clinical recommendation for radiotherapy to the primary or a metastatic lesion had been made.
* Must be able to provide informed consent.

Exclusion Criteria:

* No prior radiation to the area planned for radiotherapy
* Active invasive cancer other than pancreatic adenocarcinoma. Non-melanoma skin cancer, superficial cervical or bladder cancer and prostate cancer with PSA level < 1.0 are not excluded.
* Known HIV, HCV and/or HBV positive (by patient report/medical record)
* Patients with ongoing or active infection
* Planned concurrent treatment with systemic high dose corticosteroids.
* Received an anticancer treatment (systemic therapy or radiation therapy)within 21 days prior to enrollment.
* Immunotherapy (e.g. monoclonal antibodies)within 21 days prior to enrollment.
* Immunosuppressive therapies (e.g. steroids, cyclosporine) are not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Ben-Josef, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: In this trial, we will deliver low-dose (8Gy in a single fraction) radiotherapy (SBRT or any other acceptable delivery method as determined by the treating physician) for palliation of symptoms in patients in whom it is clinically indicated. This dose is far lower than what has been used in the definitive settings described above. This is a safe dose, and is entirely consistent with the dose range used for routine palliation. Therefore, this trial does not involve an experimental intervention; the research aspect of this protocol is the evaluation of the immune response to clinically indicated palliative radiotherapy.
  Radiation therapy
Period: Overall Study
Arm/Group | Single Arm
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (17.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=4)
Death NOS (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes